CLINICAL TRIAL: NCT01381107
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating Safety and Tolerability of ALKS 33-BUP Administration in Subjects With Major Depressive Disorder (MDD)
Brief Title: ALK33BUP-201: Safety and Tolerability Study of ALKS 33-BUP (ALKS 5461) Administration in Subjects With MDD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: ALK33BUP-201
Record Dates: First submitted 2011-06-16; First posted 2011-06-27 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — ALKS 5461

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALKS 5461 (ALKS 33 and buprenorphine) (Experimental)
  Interventions: Drug: ALKS 5461
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALKS 5461 — Sublingual administration once daily for 7 consecutive days.
  Arms: ALKS 5461 (ALKS 33 and buprenorphine)
Drug: Placebo — Sublingual administration once daily for 7 consecutive days.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel, multiple dose study designed to evaluate the safety and tolerability of the co-formulation of ALKS 33 with buprenorphine (ALKS 5461) in subjects with Major Depressive Disorder (MDD) who are inadequately/partially responding to current treatment with a stable dose of a serotonin-selective reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 18 and 65 years of age, inclusive.
* Meet Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) criteria for MDD.
* Current episode lasting ≥8 weeks prior to screening with an inadequate/partial response to an adequate trial (defined as at least 8 weeks) of a stable dose of an SSRI or SNRI. Inadequate/partial response is defined as:

  1. A Hamilton Depression Rating Scale total score (HAM-D17) ≥14, and
  2. Less than 50% reduction in depressive symptom severity on the Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (ATRQ), and
  3. Clinical Global Impression - Severity (CGI-S) score of ≥3.

Exclusion Criteria:

* Axis I diagnosis of delirium, dementia, amnestic or other cognitive disorder, schizophrenia or other psychotic disorder, bipolar I or II disorder, eating disorder, obsessive-compulsive disorder, panic disorder, or posttraumatic stress disorder.
* A clinically significant current Axis II diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal, or histrionic personality disorder.
* Experiencing hallucinations, delusions, or any psychotic symptomatology in the current episode.
* The use of inducers or inhibitors of cytochrome P450 (CYP) 3A4 (prescription medications, over-the-counter [OTC] medications, or dietary supplements) within 30 days before dosing.
* Have received electroconvulsive therapy during the current MDD episode.
* Pose current suicide risk as confirmed by the Columbia Suicide Severity Rating Scale (C SSRS).
* History of intolerance or hypersensitivity to buprenorphine.
* History of allergy or hypersensitivity to opioid antagonists (eg, naltrexone, naloxone) or quinine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The number and percent of subjects with treatment-emergent adverse events following sublingual administration of ALKS 33 and buprenorphine co-formulation (ALKS 5461) | 7 days
  Measured over a range of dose levels in subjects with inadequate/partial response to antidepressant therapy during the current episode of MDD.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Leigh-Pemberton, M.D., Study Director — Medical Director
Locations (2):
- United States (2):
  - Comprehensive NeuroScience, Inc., St. Petersburg, Florida
  - Comprehensive NeuroScience, Inc., Atlanta, Georgia